CLINICAL TRIAL: NCT06932744
Title: A Randomized, Multicenter, Active-comparator Controlled, Open-label Trial to Evaluate Efficacy and Safety of MY008211A Tablets in PNH Patients Who Are Naive to Complement Inhibitor Therapy
Brief Title: Study of Safety and Efficacy of MY008211A in Paroxysmal Nocturnal Hemoglobinuria (PNH) Patients Who Are Naive to Complement Inhibitor Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wuhan Createrna Science and Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MY008211A-PNH-3-02
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Paroxysmal Nocturnal Haemoglobinuria (PNH)
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MY008211A tablets (Experimental): MY008211A tablets 400mg BID
  Interventions: Drug: MY008211A tablets
- Eculizumab (Active Comparator): Eculizumab Injection
  Interventions: Drug: Eculizumab Injection

INTERVENTIONS:
Drug: MY008211A tablets — Participants will receive MY008211A at a dose of 400 mg orally b.i.d for 24 weeks
  Arms: MY008211A tablets
Drug: Eculizumab Injection — Eculizumab Injection for 24 weeks
  Arms: Eculizumab

SUMMARY:
The main purpose of this study is to evaluate the efficacy of MY008211A compared to eculizumab in PNH patients.

DETAILED DESCRIPTION:
This is a multi-center, randomized, open-label, active comparator-controlled, parallel group study. The purpose of this study is to determine whether MY008211A compared to eculizumab is efficacious and safe for the treatment of PNH patients who were naive to complement inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants ≥ 18 years of age and BMI ≥ 18.0 kg/m2 with a diagnosis of PNH confirmed by high-sensitivity flow cytometry with clone size ≥ 10%.
2. Mean hemoglobin level <100 g/L at screening.
3. LDH > 1.5 x Upper Limit of Normal (ULN) at screening.
4. Vaccination against Neisseria meningitidis infection is required prior to the start of study treatment. If not received previously, vaccination against Streptococcus pneumoniae and Haemophilus influenzae infections should be given.

Exclusion Criteria:

1. Patients with reticulocytes <100x10^9/L; platelets <30x10^9/L; neutrophils <0.5x10^9/L.
2. History of recurrent invasive infections caused by encapsulated organisms,e.g. meningococcus or pneumococcus.
3. Known or suspected hereditary complement deficiency.
4. Previous bone marrow or hematopoietic stem cell transplantation.
5. Previous splenectomy.
6. A history of malignancy within 5 years before screening, except cured local basal cell carcinoma of the skin and carcinoma in situ of the cervix.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of Participants With Sustained Hemoglobin Levels of ≥ 120 g/L in the Absence of Red Blood Cell Transfusions | between Day 126 and Day 168
  The proportion of patients with sustained hemoglobin levels ≥ 120 g/L among those without RBC transfusion (defined as no red blood cell infusion after D14 to D168).

SECONDARY OUTCOMES:
The proportion of subjects with an increase in hemoglobin concentration ≥ 20 g/L from baseline among subjects who do not receive RBC transfusion | between Day 126 and Day 168
  Proportion of participants achieving a sustained increase from baseline in hemoglobin levels of ≥ 20 g/L assessed among those without RBC transfusion (defined as no red blood cell infusion after D14 to D168).
The proportion of patients with LDH < 1.5 ULN among those without RBC transfusion. | between Day 126 and Day 168
  The proportion of patients with hemolysis controlled (defined as LDH < 1.5 ULN) among those without RBC transfusion
Change (Expressed as Percentages) in LDH level from baseline | between Day 126 and Day 168
  Change (Expressed as Percentages) in LDH level from baseline
Change in reticulocyte count from baseline | between Day 126 and Day 168
  Change in reticulocyte count from baseline
The proportion of patients without RBC transfusion | between Day 14 and Day 168
  The proportion of patients without RBC transfusion
Change in FACIT-F score from baseline | between Day 126 and Day 168
  Change from baseline in FACIT-Fatigue scores. The FACIT-Fatigue is a 13-item questionnaire with support for its validity and reliability in PNH that assesses patient self-reported fatigue and its impact on daily activities and function. All FACIT scales are scored so that a high score is better. As each of the 13 items of the FACIT-F Scale ranges from 0-4, the range of possible scores is 0-52, with 0 being the worst possible score and 52 the best.
The Clinical BTH Rate | between Day 1 and Day 168
  The Clinical BTH Rate
The Major Adverse Vascular Events Rate | between Day 1 and Day 168
  The Major Adverse Vascular Events Rate

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences Hematology Hospital, Tianjin, Tianjin Municipality